CLINICAL TRIAL: NCT00806585
Title: A Worldwide, Multicenter, Double-Blind, Randomized, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy & Tolerability of MK0736 When Added to Ongoing Therapy With Angiotensin-Converting Enzyme Inhibitor (ACEI) or Angiotensin Receptor Blocker (ARB) in Patients With T2DM and Hypertension
Brief Title: Dose-ranging Study to Evaluate the Effectiveness and Tolerability of MK0736 in Patients With Type 2 Diabetes Mellitus (T2DM) and Hypertension (0736-007)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0736-007; MK0736-007; 2008_600
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- MK-0736 0.5 mg (Experimental): One MK-0736 0.5 mg tablet, orally, once daily for 24 weeks (Phase A). Participant will then be switched to MK-0736 8.0 mg, once daily for an additional 52 weeks (Phase B).
  Interventions: Drug: MK-0736
- MK-0736 2.0 mg (Experimental): One MK-0736 2.0 mg tablet, orally, once daily for 24 weeks (Phase A). Participant will then be switched to MK-0736 8.0 mg, once daily for 52 weeks (Phase B).
  Interventions: Drug: MK-0736
- MK-0736 8.0 mg (Experimental): One MK-0736 8.0 mg tablet, orally, once daily for 24 weeks (Phase A). Participant will continue to receive MK-0736 8.0 mg, once daily for 52 weeks (Phase B).
  Interventions: Drug: MK-0736
- HCTZ 12.5 mg → MK-0736 8.0 mg (Active Comparator): one 12.5 mg hydrochlorothiazide (HCTZ) tablet daily, orally, for 12 weeks. Participant then switched to MK-0736 8.0 mg for 12 weeks (Phase A). Participant will continue to receive MK-0736 8.0 mg, once daily for an additional 52 weeks (Phase B).
  Interventions: Drug: MK-0736; Drug: Comparator: HCTZ
- Placebo (Placebo Comparator): One placebo tablet daily, orally, for 24 weeks (Phase A). Participant will continue to receive placebo, once daily for 52 weeks (Phase B)
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK-0736
  Arms: HCTZ 12.5 mg → MK-0736 8.0 mg; MK-0736 0.5 mg; MK-0736 2.0 mg; MK-0736 8.0 mg
Drug: Comparator: Placebo
  Arms: Placebo
Drug: Comparator: HCTZ
  Arms: HCTZ 12.5 mg → MK-0736 8.0 mg

SUMMARY:
The study will assess the efficacy and tolerability of MK0736 in patients with Type 2 Diabetes Mellitus and Hypertension who are on ongoing therapy with Angiotensin-Converting Enzyme or Angiotensin Receptor Blocker. After a 3 to 5 week pre-randomization phase, patients will be randomized to either MK0736 (3 doses), placebo, or hydrochlorothiazide (HCTZ). The study will also include a 3 week, posttreatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 to 75 years of age
* Type 2 Diabetes Mellitus (Glycohemoglobin [A1CHbA1c]: 7 to 10%)
* Hypertension: Diastolic blood pressure (DBP; 85 to 99 mm Hg) and systolic blood pressure (SBP; 120 to 159 mm Hg)
* LDL-C < 140 mg/dL
* On stable treatment with an Angiotensin-Converting Enzyme Inhibitor (ACEI) or Angiotensin Receptor Blocker (ARB)

Exclusion Criteria:

* History of Type I Diabetes mellitus or ketoacidosis
* Patients taking 3 or more blood pressure lowering medications
* Have severe chronic heart failure
* History of certain diseases or conditions such as cardiac arrhythmias, heart attack, stroke, unstable angina, or decompensated vascular disease
* History of cancer within the last 5 years
* Human immunodeficiency virus (HIV) Positive
* Have received treatment with any investigational drugs within the past 30 days
* History of alcohol or drug abuse within the past 3 years
* Body Mass Index ( BMI) >= 41 kg/m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2008-12; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study terminated after participants completed a minimum of 24 weeks of the study (i.e., Phase A) due to lack of efficacy. Phase B was not conducted.
Period: Overall Study
Arm/Group | MK-0736 0.5 mg | MK-0736 2.0 mg | MK-0736 8.0 mg | HCTZ 12.5 mg → MK-0736 8.0 mg | Placebo
Started | 137 | 134 | 141 | 71 | 137
Completed | 105 | 103 | 109 | 56 | 106
Not Completed | 32 | 31 | 32 | 15 | 31
Not completed — Study terminated by Sponsor | 0 | 0 | 1 | 2 | 0
Not completed — Protocol Violation | 3 | 1 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 3 | 0 | 1
Not completed — Lost to Follow-up | 2 | 1 | 2 | 2 | 5
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 5 | 3 | 4 | 2
Not completed — Withdrawal by Subject | 10 | 8 | 9 | 3 | 11
Not completed — Completion status unknown | 15 | 14 | 12 | 4 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0736 0.5 mg | MK-0736 2.0 mg | MK-0736 8.0 mg | HCTZ 12.5 mg → MK-0736 8.0 mg | Placebo | Total
Number analyzed (Participants) | 137 | 134 | 141 | 71 | 137 | 620
Age, Continuous [Median (Full Range); unit: years] | 58.0 [37 to 75] | 60.0 [36 to 74] | 58.0 [20 to 74] | 57.0 [37 to 74] | 58.0 [30 to 75] | 58.0 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 55 | 63 | 34 | 50 | 250
  Male | 89 | 79 | 78 | 37 | 87 | 370

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure (SiDBP) at Week 12
Description: Participant remained in the sitting position for at least 5 minutes before any blood pressure readings were recorded. Systolic and diastolic blood pressures were determined by taking 6 replicate measurements obtained 1 to 2 minutes apart. First reading was discarded and the average of the last 5 measurement was recorded.
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS) Population defined as all participants who received at least 1 dose of study drug and had endpoint data (both baseline and post-randomization)
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | MK-0736 0.5 mg | MK-0736 2.0 mg | MK-0736 8.0 mg | HCTZ 12.5 mg → MK-0736 8.0 mg | Placebo
Number analyzed (Participants) | 135 | 132 | 140 | 70 | 136
mmHg | -5.8 (0.7) | -5.7 (0.7) | -6.7 (0.7) | -7.7 (1.0) | -5.6 (0.7)
Statistical Analysis 1: Comparison: MK-0736 8.0 mg vs Placebo; Test type: Superiority or Other; p = 0.253, Constrained longitudinal data analysis; Model included terms for treatment, stratification factor, time, interaction of time by stratification factor and the interaction of time by treatment; Difference in least squares means = -1.1, 95% CI 2-sided [-3.1 to 0.8]
Statistical Analysis 2: Comparison: MK-0736 2.0 mg vs Placebo; Test type: Superiority or Other; p = 0.919, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -0.1, 95% CI 2-sided [-2.1 to 1.9]
Statistical Analysis 3: Comparison: MK-0736 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.829, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -0.2, 95% CI 2-sided [-2.2 to 1.8]
Statistical Analysis 4: Comparison: HCTZ 12.5 mg → MK-0736 8.0 mg vs Placebo; Test type: Superiority or Other; p = 0.074, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -2.1, 95% CI 2-sided [-4.5 to 0.2]
Statistical Analysis 5: Comparison: MK-0736 8.0 mg vs HCTZ 12.5 mg → MK-0736 8.0 mg; Test type: Superiority or Other; p = 0.393, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = 1.0, 95% CI 2-sided [-1.3 to 3.3]
Statistical Analysis 6: Comparison: MK-0736 2.0 mg vs HCTZ 12.5 mg → MK-0736 8.0 mg; Test type: Superiority or Other; p = 0.088, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = 2.0, 95% CI 2-sided [-0.3 to 4.4]
Statistical Analysis 7: Comparison: MK-0736 0.5 mg vs HCTZ 12.5 mg → MK-0736 8.0 mg; Test type: Superiority or Other; p = 0.108, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = 1.9, 95% CI 2-sided [-0.4 to 4.3]

2. Primary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SiSBP) at Week 12
Description: Participant remained in the sitting position for at least 5 minutes before any blood pressure readings were recorded. Systolic and diastolic blood pressures were determined by taking 6 replicate measurements obtained 1 to 2 minutes apart. First reading was discarded and the average the last 5 measurement was recorded.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | MK-0736 0.5 mg | MK-0736 2.0 mg | MK-0736 8.0 mg | HCTZ 12.5 mg → MK-0736 8.0 mg | Placebo
Number analyzed (Participants) | 135 | 132 | 140 | 70 | 136
mmHg | -5.7 (1.1) | -7.2 (1.1) | -6.3 (1.1) | -12.4 (1.5) | -5.4 (1.2)
Statistical Analysis 1: Comparison: MK-0736 8.0 mg vs Placebo; Test type: Superiority or Other; p = 0.543, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -0.9, 95% CI 2-sided [-4.0 to 2.1]
Statistical Analysis 2: Comparison: MK-0736 2.0 mg vs Placebo; Test type: Superiority or Other; p = 0.246, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -1.8, 95% CI 2-sided [-4.9 to 1.3]
Statistical Analysis 3: Comparison: MK-0736 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.821, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -0.4, 95% CI 2-sided [-3.5 to 2.7]
Statistical Analysis 4: Comparison: HCTZ 12.5 mg → MK-0736 8.0 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -7.0, 95% CI 2-sided [-10.7 to -3.3]
Statistical Analysis 5: Comparison: MK-0736 8.0 mg vs HCTZ 12.5 mg → MK-0736 8.0 mg; Test type: Superiority or Other; p = 0.001, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = 6.1, 95% CI 2-sided [2.4 to 9.8]
Statistical Analysis 6: Comparison: MK-0736 2.0 mg vs HCTZ 12.5 mg → MK-0736 8.0 mg; Test type: Superiority or Other; p = 0.006, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = 5.2, 95% CI 2-sided [1.5 to 8.9]
Statistical Analysis 7: Comparison: MK-0736 0.5 mg vs HCTZ 12.5 mg → MK-0736 8.0 mg; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = 6.7, 95% CI 2-sided [3.0 to 10.4]

3. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: LDL-C calculated by the method of Friedewald equation at baseline and after 12 weeks of study drug administration
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage Change
Arm/Group | MK-0736 0.5 mg | MK-0736 2.0 mg | MK-0736 8.0 mg | HCTZ 12.5 mg → MK-0736 8.0 mg | Placebo
Number analyzed (Participants) | 135 | 132 | 138 | 70 | 136
Percentage Change | 1.1 (2.3) | 3.9 (2.5) | 0.6 (2.5) | 2.8 (3.5) | 2.0 (2.5)
Statistical Analysis 1: Comparison: MK-0736 8.0 mg vs Placebo; Test type: Superiority or Other; p = 0.684, ANCOVA; Fixed effects for treatment baseline, stratification, time, interaction of time by stratification and treatments factors and a random subject effect; Difference in least squares means = -1.4, 95% CI 2-sided [-8.3 to 5.5]
Statistical Analysis 2: Comparison: MK-0736 2.0 mg vs Placebo; Test type: Superiority or Other; p = 0.597, ANCOVA; [statistical method as in outcome 3, analysis 1]; Difference in least squares means = 1.8, 95% CI 2-sided [-5.0 to 8.7]
Statistical Analysis 3: Comparison: MK-0736 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.793, ANCOVA; [statistical method as in outcome 3, analysis 1]; Difference in least squares means = -0.9, 95% CI 2-sided [-7.6 to 5.8]
Statistical Analysis 4: Comparison: HCTZ 12.5 mg → MK-0736 8.0 mg vs Placebo; Test type: Superiority or Other; p = 0.854, ANCOVA; [statistical method as in outcome 3, analysis 1]; Difference in least squares means = 0.8, 95% CI 2-sided [-7.6 to 9.2]

4. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: Fasting weight was assessed at baseline and after 24 weeks of study drug administration and was measured after voiding, with shoes and socks off, wearing clinic gown to reduce variability and maintain consistency. Same standardized digital scale was used throughout the study.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | MK-0736 0.5 mg | MK-0736 2.0 mg | MK-0736 8.0 mg | HCTZ 12.5 mg → MK-0736 8.0 mg | Placebo
Number analyzed (Participants) | 135 | 132 | 140 | 70 | 136
kg | -0.7 (0.5) | -1.4 (0.5) | -1.3 (0.5) | -1.6 (0.7) | 0.6 (0.5)
Statistical Analysis 1: Comparison: MK-0736 8.0 mg vs Placebo; Test type: Superiority or Other; p = 0.006, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -1.9, 95% CI 2-sided [-3.2 to -0.5]
Statistical Analysis 2: Comparison: MK-0736 2.0 mg vs Placebo; Test type: Superiority or Other; p = 0.004, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -2.0, 95% CI 2-sided [-3.3 to -0.6]
Statistical Analysis 3: Comparison: MK-0736 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.066, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Diffference in least squares means = -1.3, 95% CI 2-sided [-2.6 to 0.1]
Statistical Analysis 4: Comparison: HCTZ 12.5 mg → MK-0736 8.0 mg vs Placebo; Test type: Superiority or Other; p = 0.008, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -2.2, 95% CI 2-sided [-3.7 to -0.6]

5. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 24
Description: HbA1c reported as a % and was measured at baseline and after 24 weeks of study drug administration
Time Frame: Baseline and Week 24
Population: Full Analysis Set (FAS) Population defined as all participants who received at least 1 dose of study drug and did not lack of any endpoint data (both baseline and post-randomization)
Measure: Least Squares Mean (Standard Error); unit: Percentage Change
Arm/Group | MK-0736 0.5 mg | MK-0736 2.0 mg | MK-0736 8.0 mg | HCTZ 12.5 mg → MK-0736 8.0 mg | Placebo
Number analyzed (Participants) | 135 | 132 | 140 | 70 | 136
Percentage Change | -0.10 (0.09) | -0.16 (0.10) | -0.06 (0.09) | -0.20 (0.13) | 0.13 (0.10)
Statistical Analysis 1: Comparison: MK-0736 8.0 mg vs Placebo; Test type: Superiority or Other; p = 0.152, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -0.18, 95% CI 2-sided [-0.44 to 0.07]
Statistical Analysis 2: Comparison: MK-0736 2.0 mg vs Placebo; Test type: Superiority or Other; p = 0.035, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least sqaures means = -0.28, 95% CI 2-sided [-0.54 to -0.02]
Statistical Analysis 3: Comparison: MK-0736 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.095, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -0.22, 95% CI 2-sided [-0.48 to 0.04]
Statistical Analysis 4: Comparison: HCTZ 12.5 mg → MK-0736 8.0 mg vs Placebo; Test type: Superiority or Other; p = 0.045, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -0.32, 95% CI 2-sided [-0.63 to -0.01]

ADVERSE EVENTS:
Time Frame: 76 weeks
Description: All Randomized Participants. Adverse events were reported for Phase A only (24 weeks). Phase B (52 weeks) was not completed.
Arm/Group | MK-0736 0.5 mg | MK-0736 2.0 mg | MK-0736 8.0 mg | HCTZ 12.5 mg → MK-0736 8.0 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 9/137 | 7/134 | 6/141 | 0/71 | 5/137
Other Adverse Events (participants affected / at risk) | 46/137 | 54/134 | 54/141 | 25/71 | 43/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0736 0.5 mg (N=137) | MK-0736 2.0 mg (N=134) | MK-0736 8.0 mg (N=141) | HCTZ 12.5 mg → MK-0736 8.0 mg (N=71) | Placebo (N=137)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresis cranial nerve (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0736 0.5 mg (N=137) | MK-0736 2.0 mg (N=134) | MK-0736 8.0 mg (N=141) | HCTZ 12.5 mg → MK-0736 8.0 mg (N=71) | Placebo (N=137)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 8 (10) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 8 (9) | 3 (4) | 2 (2) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 8 (12) | 10 (17) | 7 (7) | 4 (5) | 7 (9)
Low density lipoprotein increased (Investigations) | 9 (10) | 10 (10) | 9 (9) | 5 (5) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 24 (118) | 24 (79) | 28 (91) | 9 (91) | 27 (197)
Headache (Nervous system disorders) | 4 (5) | 8 (12) | 10 (13) | 4 (8) | 8 (8)
Hypertension (Vascular disorders) | 4 (5) | 4 (4) | 9 (9) | 1 (1) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.